CLINICAL TRIAL: NCT02243722
Title: Establish Comprehensive Quantitative Measurements of Laryngeal Sensorimotor Functions and Evaluating the Grade of Phonation and Swallowing Impairment
Brief Title: Establish Quantitative Measurements of Laryngeal Sensorimotor Functions and Evaluating the Grade of Phonation and Swallowing Impairment
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 102-5333A3
Record Dates: First submitted 2014-09-16; First posted 2014-09-18 (Estimated); Last update posted 2014-09-18 (Estimated); Status verified 2014-02

CONDITIONS: Unilateral Vocal Cord Paralysis
Keywords: laryngeal electromyography; intrinsic laryngeal muscles; recurrent laryngeal nerve; superior laryngeal nerve; laryngeal sensation; tone language
MeSH Terms: conditions — Vocal Cord Paralysis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Larynx pharynx and Esophagus Ca with VCP: The cases of laryngopharyngeal and esophageal cancer with endoscopic characters of vocal fold motion impairment (paralysis or fixation)

SUMMARY:
Laryngeal motor and sensory nerve dysfunction may cause phonation and swallowing disturbance, which often happens after the treatment for laryngopharyngeal and esophageal cancer and may induce fatal complications such as aspiration pneumonia. By the conventional examinations, the tiny sensory or motor changes are hard to be detected before complete vocal paralysis. It is utmost important to establish a comprehensive quantitative method which is sensitive enough to evaluate the neuromuscular functions. The present project will evaluate the laryngeal nerve function by quantitative laryngeal electromyography, which was developed by the research team, and another novel examination technique, mucosal membrane sensation test. The comprehensive method is expected to grade the laryngeal nerve injuries quantitatively before the significant symptoms or complications and can also help to evaluate the treatment effect from medicine, rehabilitation or surgery.

ELIGIBILITY:
Inclusion Criteria:

* Patients with laryngopharyngeal or esophageal cancer who have taken active therapy and are not neck tissue damage.
* Patients with clear conscious and stable mental status

Exclusion Criteria:

* Patients who cannot sit for longer than 30 minutes or received other vocal cord treatments before the selection
* Pregnant and breastfeeding women
* Patients with communication disorder

Ages: 20 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients from a tertian referral medical center.
Sampling Method: Non-Probability Sample
Enrollment: 70 (Estimated)
Dates: Start 2014-07; Primary Completion 2016-08 (Estimated); Study Completion 2016-11 (Estimated)

PRIMARY OUTCOMES:
Fiberoptic endoscopic evaluation of swallowing (FEES) | Baseline:Within 3-6 months after synptom occurs
  Swallowing evaluation
Laryngo-pharyngeal mucosa sensation test | Baseline:Within 3-6 months after synptom occurs
  There were four probes of different diameters that similar to the Von Frey filament were prepared for the examination. The diameters were 0.07mm, 0.15mm.0.2 mm and 0.3 mm. The mono-filament nylon probe was placed and contact with the tip and arytenoid mucosa.

SECONDARY OUTCOMES:
laryngeal electromyography | Baseline:Within 3-6 months after synptom occurs
laboratory voice analysis | Baseline:Within 3-6 months after synptom occurs
  fundamental frequency, Jitter (perturbation of frequency), Shimmer (perturbation of amplitude), harmonic-to-noise ratio (HN), and s/z ratio (SZ) .
voice range profile | Baseline:Within 3-6 months after synptom occurs
  The voice will be analyzed by computerized software. The extreme lowest and highest notes of frequencies production and the amplitude will be recorded and a voice map will be made as a plot of sound pressure level versus F0.
Voice Handicap Index (VHI) | Baseline:Within 3-6 months after synptom occurs
  Voice-related questionnaire The Voice Handicap Index (VHI) is a 30-item instrument developed by Jacobson et al. as a self-measure the psychosocial handicapping effects of voice disorders. The questionnaire consists of three sub scales: emotional, physical and functional with 10 items from each scale. It has been translated into traditional Chinese and validated. All individuals will be asked to response for the questionnaire.
Disease related life quality assessment: FACT-H&N, FACT-E | Baseline:Within 3-6 months after synptom occurs
  Functional Assessment of Cancer Therapy-Head and Neck (FACT-H&N) and FACT-E (esophagus) are self -report questionnaires with a Likert-type response set, ranging from "not at all" to "very much". FACT-G (general) is a 27-items scale measures four QOL (quality of life) domains including Physical Well-Being, Social/Family Well-Being, Emotional Well-Being and Functional Well-Being. In FACT-H&N, there are 11 additional specific questions for head and neck cancers while 17 additional items for esophageal cancers in FACT-E. The specific questionnaires will be provided to patients according to individual diseases. The traditional Chinese (Mandarin) version has been validated and proved to be useful in previous report. We have received the licensing agreement from the institute (FACIT) for using the questionnaires on the project.

CONTACTS AND LOCATIONS:
Overall Officials: Tuan-Jen Fang, MD, Principal Investigator — Chang Gung Memorial Hospital
Locations (1):
- Chang Gung Memorial Hospital, Taoyuan District, Taiwan